CLINICAL TRIAL: NCT03830008
Title: Scaling-up Psychological Interventions With Syrian Refugees in Switzerland
Acronym: STRENGTHS_CH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-2017-01175
Record Dates: First submitted 2019-01-07; First posted 2019-02-05 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Distress; PTSD; Anxiety; Depression; Trauma; Functional Disabilities; Common Mental Health Problems
Keywords: Problem Management Plus; Distress; Mental Health Care; Low-intensity; Refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The exploratory RCT will inform us about the feasibility, safety, and delivery of the intervention; this will identify issues around its training, supervision and outcome measures.
  After the baseline assessment, sixty participants (N = 60) will be involved in the exploratory RCT (assigned to either the PM+ intervention (n=30) or the ETAU control condition (n=30)). The investigators intend to deliver the intervention to 30 participants, allowing us to test the feasibility and acceptability of the intervention in the proposed setting and inform the sample size for a future definitive trial.
Who Masked: Outcomes Assessor
Masking Description: All instruments and questions will be administered using tablets by trained research staff blind to the allocation status of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment As Usual (ETAU) (No Intervention): The control group will receive enhanced treatment as usual (ETAU). ETAU means that the research team will advise the participants to contact their doctor in case of physical or mental health problems. Moreover, the research team will hand over the list with the general practitioners (GP) in the neighborhood of the participant and the written information (official booklet) about the operating of the Swiss health care system. Adequate treatment will be provided by this physician, usually, a general practitioner who acts as a gate-keeper (an asylum seeker or refugee has to go first to his/her assigned GP in order to get access to the health care system).
- Problem Management Plus (Experimental): PM+ is a new, brief, psychological intervention program based on Cognitive Behaviour Therapy (CBT) techniques that are empirically supported and formally recommended by the WHO. The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, facing fears, and accessing social support. These elements have been recommended in recent WHO guidelines.
  Interventions: Behavioral: Problem Management Plus

INTERVENTIONS:
Behavioral: Problem Management Plus — PM+ is a new, brief, psychological intervention program based on CBT techniques that are empirically supported and formally recommended by the WHO. The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, facing fears, and accessing social support. These elements have been recommended in recent WHO guidelines.
  Arms: Problem Management Plus

SUMMARY:
The current refugee crisis across the Middle East and Europe has large effects on individual refugees' psychological well-being, as well as on the healthcare systems of countries hosting refugees. For example, in Switzerland patients sometimes have to wait up to 12 months for the specific psychological treatment due to a lack of specialists. To address this problem the WHO has developed Problem Management Plus (PM+), a brief (five sessions), low-intensity psychological intervention, delivered by paraprofessionals, that addresses common mental disorders in people in communities affected by adversity. The feasibility of PM+ has never been examined in Switzerland before, this is the aim of the current pilot study.

DETAILED DESCRIPTION:
Recent crises in the Middle East, most notably in Syria, have resulted in an unprecedented increase in the worldwide number of refugees and asylum seekers. Switzerland (CH) is strongly affected by this crisis too. Eight percent of asylum requests in 2016 were made by people from Syria (2015: 12 %). More than 7'000 asylum seekers from Syria entered CH over the last two years. Due to the ongoing war in this region, it is unlikely that this kind of migration and flight will stop. Notably, 50% of the refugee population are children and adolescents.

Refugees have typically been exposed to multiple stressors related to war and displacement including loss of family members, destruction of homes and livelihoods and human rights violations such as sexual violence or torture. They have often undertaken a risky and stressful flight leaving their homes for an unknown future. Accordingly, studies consistently show that refugees are at considerable risk of developing common mental disorders, including depression, anxiety, posttraumatic stress disorder (PTSD) and related somatic health symptoms. Recent WHO projections suggest that approximately 15-20% of Syrian refugees will develop some type of mental health problem and therefore represent an enormous public mental health challenge.

According to the UNHCR, 86% of all displaced persons remain in conflict or neighboring countries where appropriate health care is mostly not available. But also Western health systems are often unable to appropriately cover the needs of this particularly vulnerable population regarding prevention and treatment of mental health problems. As a response to this situation, the WHO developed the low-intensity Problem Management Plus (PM+) programs, a new generation of shorter, less expensive and trans-diagnostic (i.e., not specifically aimed at treating a certain mental disorder) programs to reduce common mental health symptoms and improve psychosocial functioning. PM+ is based on the WHO treatment guidelines for conditions related to stress. PM+ is a 5-sessions intervention aimed at reducing symptoms of depression, anxiety, PTSD, and related conditions, is delivered by trained non-specialized workers or lay people, and is available in individual and group delivery formats for both children and adults. It comprises evidence-based techniques of (a) problem solving, (b) stress management, (c) behavioral activation, and (d) accessing social support. PM+ has been successfully implemented in Kenya and Pakistan.

The STRENGTHS (Syrian REfuGees MeNTal HealTH Care Systems) study aims at evaluating the effectiveness and implementation of PM+ with Syrian refugees in different settings in low- and high-resource countries. The study consortium includes international experts in the domains of trauma and public mental health as well as representatives of WHO and UNHCR. The Zürich study site has been consigned to examine PM+ with adult refugees in an individual treatment setting in Switzerland. At the same time, similar studies in other countries will be undertaken. Despite the objective of these studies to implement and evaluate the effectiveness of PM+ in refugees, each research institution acts independently. Moreover, the other studies will be completed in different treatment settings - i.e., in children and adolescents (Lebanon), in groups (Turkey and Netherlands), and internet-delivered PM+ (Germany and Egypt).

To date, the feasibility of PM+ has not been investigated in a highly industrialized country, such as Switzerland.

In the present study, the investigators will evaluate the feasibility of PM+ in Syrian refugees in Switzerland.

This research entails single-blind randomized controlled trial.

The amendment was secured by December 2018. Trainers, assessors, supervisors and helpers are already identified, recruited an trained.

After the approval, the first participants will be identified, invited to screening and if they fulfill the criteria they will be invited to participate in the pilot study. The pilot study will end by the end of 2019. After the pilot study the results will be evaluated, analyzed and integrated in the planning of the definitive randomized controlled trial (RCT) (next study, not the part of current registration).

ELIGIBILITY:
Inclusion Criteria:

* Male and female Syrian refugees or asylum seekers who entered Switzerland after the beginning of Syrian Civil War in March 2011
* ≥ 18 years of age
* Arabic-speaking
* Signed Informed Consent after being informed
* Increased psychological distress (K10 > 15)
* Reduced psychological functioning (WHODAS 2.0 > 16)

Exclusion Criteria:

* Inability to follow the procedures of the study
* Previous enrolment into the current study
* Previous or currently enrolment of a family member into the current study
* Participants under tutelage
* Acute or severe psychiatric (e.g. schizophrenia) or neurological illness (e.g. dementia)
* Imminent suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Verification procedure to the measurement in psychological distress at baseline assessment | baseline assessment (before PM+)
  measured by the Hopkins Symptom Checklist (HSCL-25)
Verification procedure to the measurement in psychological distress after PM+ intervention or ETAU | post-assessment baseline (after PM+/ETAU)
  measured by the Hopkins Symptom Checklist (HSCL-25)
Verification procedure to the measurement in psychological distress 3 months after PM+ intervention or ETAU | 3-months follow-up (after PM+/ETAU)
  measured by the Hopkins Symptom Checklist (HSCL-25)

SECONDARY OUTCOMES:
Verification procedure to the measurement of symptoms of posttraumatic stress disorder at baseline assessment | baseline assessment (before PM+)
  measured using the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5)
Verification procedure to the measurement of symptoms of posttraumatic stress disorder after PM+ intervention or ETAU | post-assessment baseline (after PM+/ETAU)
  measured using the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5)
Verification procedure to the measurement of symptoms of posttraumatic stress disorder 3 months after PM+ intervention or ETAU | 3-months follow-up (after PM+/ETAU)
  measured using the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5)
Verification procedure to the measurement of functional disability at screening | screening (before PM+)
  assessed by the WHODAS 2.0 (WHO Disability Assessment Schedule 2.0)
Verification procedure to the measurement of functional disability after PM+ intervention or ETAU | post-assessment baseline (after PM+/ETAU)
  assessed by the WHODAS 2.0 (WHO Disability Assessment Schedule 2.0)
Verification procedure to the measurement of functional disability 3 months after PM+ intervention or ETAU | 3-months follow-up (after PM+/ETAU)
  assessed by the WHODAS 2.0 (WHO Disability Assessment Schedule 2.0)
Feasibility of PM+ by the number of dropouts | screening (before PM+)
  Monitoring of the dropouts by number of patients
Feasibility of PM+ by the number of dropouts | baseline assessment (before PM+)
  Monitoring of the dropouts by number of patients
Feasibility of PM+ by the number of dropouts | post-assessment baseline (after PM+/ETAU)
  Monitoring of the dropouts by number of patients
Feasibility of PM+ by the number of dropouts | 3-months follow-up (after PM+/ETAU)
  Monitoring of the dropouts by number of patients
Feasibility of PM+ by feedbacks regarding the understanding of intervention and measurements instruments | screening (before PM+)
  Monitoring of wrong understanding or wrong translation (by number of patients and the scope of the feedback)
Feasibility of PM+ by feedbacks regarding the understanding of intervention and measurements instruments | baseline assessment (before PM+)
  Monitoring of wrong understanding or wrong translation (by number of patients and the scope of the feedback)
Feasibility of PM+ by feedbacks regarding the understanding of intervention and measurements instruments | post-assessment baseline (after PM+/ETAU)
  Monitoring of wrong understanding or wrong translation (by number of patients and the scope of the feedback)
Feasibility of PM+ by feedbacks regarding the understanding of intervention and measurements instruments | 3-months follow-up (after PM+/ETAU)
  Monitoring of wrong understanding or wrong translation (by number of patients and the scope of the feedback)

OTHER OUTCOMES:
Verification procedure to the measurement of change in response to therapy at baseline | baseline assessment (before PM+)
  patient-generated outcome measure by the Psychological Outcomes Profiles (PSYCHLOPS) scale [PSYCHLOPS has questions on Problems, Function and Wellbeing. Participants are asked to describe their main Problem or Problems and how this affects them (Function). Responses to all questions are scored [likert-scale 0 to 5 from "severely affected" to "not at all affected"); it is a highly sensitive measure of change during the course of psychotherapeutic interventions.]
Verification procedure to the measurement of change in response to therapy at post-assessment | post-assessment baseline (after PM+/ETAU)
  patient-generated outcome measure by the Psychological Outcomes Profiles (PSYCHLOPS) scale [PSYCHLOPS has questions on Problems, Function and Wellbeing. Participants are asked to describe their main Problem or Problems and how this affects them (Function). Responses to all questions are scored [likert-scale 0 to 5 from "severely affected" to "not at all affected"); it is a highly sensitive measure of change during the course of psychotherapeutic interventions.]
Verification procedure to the measurement of change in response to therapy 3 months after | 3-months follow-up (after PM+/ETAU)
  patient-generated outcome measure by the Psychological Outcomes Profiles (PSYCHLOPS) scale [PSYCHLOPS has questions on Problems, Function and Wellbeing. Participants are asked to describe their main Problem or Problems and how this affects them (Function). Responses to all questions are scored [likert-scale 0 to 5 from "severely affected" to "not at all affected"); it is a highly sensitive measure of change during the course of psychotherapeutic interventions.]
Post-migration stressors at baseline | baseline assessment (before PM+)
  will be assessed using a version of the Post-Migration Living Difficulties Checklist (PMLDC)
Post-migration stressors at post-assessment | post-assessment baseline (after PM+/ETAU)
  will be assessed using a version of the Post-Migration Living Difficulties Checklist (PMLDC)
Post-migration stressors 3 months after | 3-months follow-up (after PM+/ETAU)
  will be assessed using a version of the Post-Migration Living Difficulties Checklist (PMLDC)
Previous exposure to traumatic events | baseline
  assessed using the Traumatic Events (TE) - a combination of two standardized questionnaires, namely the Life Events Checklist (LEC) (Weathers et al., 2013) and the Harvard Trauma Questionnaire (HTQ) (Mollica et al., 1992). HTQ consists of 3 sections with 48 questions. LEC consists of 17 question. Single questions from HTQ (Section 1) and LEC are summarized to the sequence of 27 questions (about experienced trauma or adversities with yes/no answer format). The number of positive answers is the outcome value.
Access to Health Care Services (AHCS) | baseline assessment (before PM+)
  The set of question regarding previous contact with the mental health care services and the previous experiences regarding the utilization of any forms of mental support
Medical service utilization of people with mental disorders at baseline | baseline assessment (before PM+)
  accessed using the Client Service Receipt Inventory (CSRI) as the basis for calculating the costs of care for mental health cost-effectiveness research
Medical service utilization of people with mental disorders at post-assessment | post-assessment baseline (after PM+/ETAU)
  accessed using the Client Service Receipt Inventory (CSRI) as the basis for calculating the costs of care for mental health cost-effectiveness research
Medical service utilization of people with mental disorders at post-assessment 3 months after | 3-months follow-up (after PM+/ETAU)
  accessed using the Client Service Receipt Inventory (CSRI) as the basis for calculating the costs of care for mental health cost-effectiveness research

CONTACTS AND LOCATIONS:
Overall Officials: Naser Morina, PhD, Principal Investigator — University Hospital Zurich / University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sijbrandij M, Acarturk C, Bird M, Bryant RA, Burchert S, Carswell K, de Jong J, Dinesen C, Dawson KS, El Chammay R, van Ittersum L, Jordans M, Knaevelsrud C, McDaid D, Miller K, Morina N, Park AL, Roberts B, van Son Y, Sondorp E, Pfaltz MC, Ruttenberg L, Schick M, Schnyder U, van Ommeren M, Ventevogel P, Weissbecker I, Weitz E, Wiedemann N, Whitney C, Cuijpers P. Strengthening mental health care systems for Syrian refugees in Europe and the Middle East: integrating scalable psychological interventions in eight countries. Eur J Psychotraumatol. 2017 Nov 7;8(sup2):1388102. doi: 10.1080/20008198.2017.1388102. eCollection 2017. PMID 29163867
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Hassan, G., Kirmayer, L. J., Mekki-Berrada, A., Quosh, C., el Chammay, R., Deville-Stoetzel, J., . . . Coutts, A. (2015). Culture, context and the mental health and psychosocial wellbeing of Syrians: a review for mental health and psychosocial support staff working with Syrians affected by armed conflict. Geneva: UNHCR.
- [Background] Guidelines for the Management of Conditions Specifically Related to Stress. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK159725/ PMID 24049868
- [Background] Rahman A, Riaz N, Dawson KS, Usman Hamdani S, Chiumento A, Sijbrandij M, Minhas F, Bryant RA, Saeed K, van Ommeren M, Farooq S. Problem Management Plus (PM+): pilot trial of a WHO transdiagnostic psychological intervention in conflict-affected Pakistan. World Psychiatry. 2016 Jun;15(2):182-3. doi: 10.1002/wps.20312. No abstract available. PMID 27265713
- [Background] Steel Z, Chey T, Silove D, Marnane C, Bryant RA, van Ommeren M. Association of torture and other potentially traumatic events with mental health outcomes among populations exposed to mass conflict and displacement: a systematic review and meta-analysis. JAMA. 2009 Aug 5;302(5):537-49. doi: 10.1001/jama.2009.1132. PMID 19654388
- [Background] Dua T, Barbui C, Clark N, Fleischmann A, Poznyak V, van Ommeren M, Yasamy MT, Ayuso-Mateos JL, Birbeck GL, Drummond C, Freeman M, Giannakopoulos P, Levav I, Obot IS, Omigbodun O, Patel V, Phillips M, Prince M, Rahimi-Movaghar A, Rahman A, Sander JW, Saunders JB, Servili C, Rangaswamy T, Unutzer J, Ventevogel P, Vijayakumar L, Thornicroft G, Saxena S. Evidence-based guidelines for mental, neurological, and substance use disorders in low- and middle-income countries: summary of WHO recommendations. PLoS Med. 2011 Nov;8(11):e1001122. doi: 10.1371/journal.pmed.1001122. Epub 2011 Nov 15. PMID 22110406
- [Background] Tol WA, Barbui C, van Ommeren M. Management of acute stress, PTSD, and bereavement: WHO recommendations. JAMA. 2013 Aug 7;310(5):477-8. doi: 10.1001/jama.2013.166723. No abstract available. PMID 23925613
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP): Version 2.0. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK390828/ PMID 27786430
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P., Marx, B., & Schnurr, P. (2013). The ptsd checklist for dsm-5 (pcl-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Mollica RF, Caspi-Yavin Y, Bollini P, Truong T, Tor S, Lavelle J. The Harvard Trauma Questionnaire. Validating a cross-cultural instrument for measuring torture, trauma, and posttraumatic stress disorder in Indochinese refugees. J Nerv Ment Dis. 1992 Feb;180(2):111-6. PMID 1737972